CLINICAL TRIAL: NCT05749081
Title: Lacidophilin Tablets in Combination With Vonorazan and Amoxicillin Dual Therapy for Eradicating Helicobacter Pylori Infection: a Prospective, Multi-centers, Superiority, Double-blind, Randomized Clinical Study
Brief Title: Helicobacter Pylori and Lacidophilin Tablets in Combination With Vonorazan Dual Therapy
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Lingyu Luo, Professor, The First Affiliated Hospital of Nanchang University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Hp therapy of FirstNanchangU
Record Dates: First submitted 2023-02-18; First posted 2023-03-01 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; vonoprazan; Lacidophilin Tablets; amoxicillin; eradication

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lacidophilin tablets group (Experimental): 2400mg lacidophilin tablets three times daily,1000mg amoxicillin capsules three times daily and 20mg vonoprazan Fumarate Tablets twice daily for 10 days
  Interventions: Drug: Lacidophilin tablets in combination with vonorazan dual therapy
- Placebo group (Placebo Comparator): 2400mg placebo three times daily,1000mg amoxicillin capsules three times daily and 20mg vonoprazan Fumarate Tablets twice daily for 10 days
  Interventions: Drug: Placebo in combination with vonorazan dual therapy

INTERVENTIONS:
Drug: Lacidophilin tablets in combination with vonorazan dual therapy — 2400mg lacidophilin tablets three times daily,1000mg amoxicillin capsules three times daily and 20mg vonoprazan Fumarate Tablets twice daily for 10 days
  Arms: Lacidophilin tablets group
Drug: Placebo in combination with vonorazan dual therapy — 2400mg placebo three times daily,1000mg amoxicillin capsules three times daily and 20mg vonoprazan Fumarate Tablets twice daily for 10 days
  Arms: Placebo group

SUMMARY:
Our previous study included 119 Helicobacter pylori(H. pylori)-infected Chinese patients without previous eradication history who were randomized to low-or high-dose amoxicillin-vonoprazan regimens consisting of amoxicillin 1 gram either b.i.d. or t.i.d plus vonoprazan 20 mg b.i.d for 7 or 10 days. Neither 7-or 10-day VA dual therapy with either b.i.d. or t.i.d. amoxicillin achieved satisfied efficacy (i.e., <90%) when given as first-line treatment for H. pylori infection. Lacidophilin tablets have been reported to increase the eradication rate of H. pylori while reducing the incidence of adverse effects.This study evaluated the efficacy and safety of lacidophilin tablets in combination with amoxicillin-vonoprazan dual therapy for 10 days as first-line treatment for H. pylori in China.

DETAILED DESCRIPTION:
This study was designed as a prospective, multi-centers, double-blind, randomized superiority clinical study and was conducted in accordance with the Declaration of Helsinki and the guidelines of the Consolidated Standards of Reporting Trials.

Consecutive H. pylori-infected subjects ages from 18 to 70 without eradication history were recruited . H. pylori infection was confirmed by immunohistochemistry or urea breath test.

The H. pylori-infected subjects were randomly assigned to receive lacidophilin tablets or placebo in combination with amoxicillin-vonoprazan dual therapy for in a 1:1 allocation ratio, a randomization list was generated using Statistical Product Service Solutions (version 25.0).

The therapy consisted of 2400mg lacidophilin tablets or placebo three times daily, 1000 mg amoxicillin capsules three times daily and 20mg vonoprazan fumarate tablets twice daily for 10 days. The shape, taste, packaging, storage method and administration method of placebo are the same as lacidophilin tablets. Participants and investigators were blinded to the allocated treatment group.

At the start, the detailed demographics and characteristics of the subjects included in this study were recorded, including sex, age, nationality, height, weight, education status, dwelling area, history of smoking and alcohol, concomitant diseases and medication history. In addition, physical examinations and assessment of vital signs were performed. Gastric antrum and body biopsy of the included subjects were obtained during the endoscopy, which were followed by culture and susceptible test of antibiotics. Fecal sample was collected before eradication.

During (or after) treatment-emergent adverse events (TEAEs) and concomitant medication were recorded throughout the study, including bloating, nausea, vomiting, abdominal pain, diarrhea, constipation, skin rash, headache, hunger sensation and others. All TEAEs were divided into mild, moderate and severe, TEAEs leading to study drug discontinuation were also recorded. Fecal sample was collected after eradication.

The confirmation of H. pylori status was evaluated by 13C-urea breath test 4-8 weeks after treatment. H. pylori status was considered as negative or positive according to the instructions of the manufacturer. Oral and fecal sample was collected at the timepoint of recheck.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive H. pylori-infected subjects ages from 18 to 70 without eradication history

Exclusion Criteria:

* allergy to amoxicillin,vonoprazan or lacidophilin tablets;
* acute upper gastrointestinal bleeding, gastric cancer or other tumors, Zollinger-Ellison syndrome, history of gastric surgery;
* gastroscopy report showing or past medical history of significant esophagogastric disease, including gastric cancer, peptic ulcer, esophagitis, esophageal erosion.
* serious illness including neurological, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, urological, endocrinological or hematological disorders;
* pregnancy or breast feeding;
* proton pump inhibitors, antibiotics and probiotics use within one month;
* not willing to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2023-05-13 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Treatment | 4-8 weeks after treatment
  The confirmation of H. pylori status was evaluated by urea breath test

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 1 day after eradication
  the frequency and severity of treatment-emergent adverse events
Compliance of Participants | 1 day after eradication
  good compliance was defined as achieving ≥80% of drugs included in the regimes and bad compliance was defined as achieving <80% drugs
Resistance of Antibiotics | before the eradication
  An E-test was used to determine the minimum inhibitory concentrations (MIC) of Amoxicillin (AMO), Metronidazole (MET), Clarithromycin (CLA), Levofloxacin (LEV) and tetracycline (TET). The Kirby-Bauer disc diffusion method (Oxoid) was used to determine the inhibition zone for Furazolidone (FUR). A strain was considered resistant if the MIC>1 mg/mL for AMO, ≥1 mg/mL for CLA, >2 mg/mL for TET, >4 mg/mL for MET, MIC >1 mg/mL for LEV and if the inhibition zone was <7 mm for FUR. H. pylori strain ATCC 43504 was included as an antibiotic susceptibility testing qualitycontrol. All antibiotic susceptibility tests were conducted at the Institute of Gastroenterology and Hepatology, First Affiliated Hospital of Nanchang University.
Alteration of Gut Microbiota | before eradication，1 day after eradication and confirmation（4-8 weeks after treatment）
  The oral and fecal samples were collected before eradication,1 day after eradication and confirmation（6-8 weeks after treatment）. Bioinformatics of gut microbiome were performed using QIIME2 with slight modification and R packages. Briefly, Non-singleton ASVs were aligned and used to construct a phylogeny with fasttree2. Alpha-diversity metrics were calculated using the ASV table in QIIME2 and visualized as box plots. ASV-level ranked abundance curves were generated to compare the richness and evenness of ASVs among samples. Beta diversity analysis was conducted to explore the structural variation of microbial communities across samples using Bray-Curtis metrics and visualized via principal coordinate analysis (PCoA). The significance of microbiota structure differences among groups was assessed by Permanova using QIIME2. Microbial functions were predicted by PICRUSt2 upon KEGG (https://www.kegg.jp/) databases.

CONTACTS AND LOCATIONS:
Overall Officials: Cong He, phD, Principal Investigator — The First Affiliated Hospital of Nanchang University
Locations (1):
- The first affiliated hospital, Jiangxi Medical College, NanChang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No